CLINICAL TRIAL: NCT00255606
Title: A Phase III Trial Comparing Docetaxel Every Third Week to Biweekly Docetaxel Monotherapy in Metastatic Hormone Refractory Prostate Cancer Patients - PROSTY Trial
Brief Title: Docetaxel and Prednisone in Treating Patients With Hormone-Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: AVENTIS-FIN-1-2003; CDR0000442891 (Registry Identifier: PDQ (Physician Data Query)); FINNISH-URO-OGS-1-2003; PROSTY-FIN-1-2003; ICORG-06-14-Prosty; EU-20891
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2010-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone

ARMS (2):
- Arm I (Experimental): Patients receive docetaxel IV over 1 hour on days 1 and 15 and oral prednisone once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: prednisone
- Arm II (Experimental): Patients receive docetaxel IV over 1 hour on day 1 and prednisone once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: prednisone

INTERVENTIONS:
Drug: docetaxel — Given in 3- or 4- week courses
Drug: prednisone — Given in 3- or 4- week courses

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known which schedule of docetaxel and prednisone is more effective in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying two different schedules of docetaxel and prednisone to compare how well they work in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the time to treatment failure in patients with hormone-refractory metastatic prostate cancer treated with two different schedules of docetaxel in combination with prednisone.

Secondary

* Compare overall survival of patients treated with these regimens.
* Compare the response rate in patients treated with these regimens.
* Compare the safety of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Compare the need for epoetin beta in patients treated with these regimens.
* Determine the effect of epoetin beta on hemoglobin response rate, transfusion rate, and quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to participating center and WHO performance status (0-1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on days 1 and 15 and oral prednisone once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive docetaxel IV over 1 hour on day 1 and prednisone once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients who experience anemia (hemoglobin < 11 g/dL) receive epoetin beta subcutaneously once weekly during chemotherapy.

Quality of life is assessed at baseline, every 6 weeks during study treatment, at completion of study treatment, and then every 2 months thereafter.

After completion of study treatment, patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 360 patients (180 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * Metastatic disease by imaging or clinical examination
* Hormone-refractory disease, defined as prostate-specific antigen (PSA) level > 10 µg/L AND rising between 2 sequential measurements
* Testosterone within castration levels by orchiectomy or medical castration comprising luteinizing hormone-releasing hormone (LHRH) analogues

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count ≥ 1,500/mm^3
* Hemoglobin ≥ 11.0 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* ALT and AST ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin normal
* Alkaline phosphatase ≤ 6 times ULN (unless due to the presence of extensive bone disease)
* No serious liver disease

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No ischemic or thromboembolic cardiac disease
* No myocardial infarction within the past 12 months
* No other serious cardiac disease

Pulmonary

* No pulmonary emboli

Immunologic

* No active infection
* No autoimmune disease, including any of the following:

  * Lupus
  * Scleroderma
  * Rheumatoid polyarthritis

Other

* No active peptic ulcer
* No unstable diabetes mellitus
* No contraindication to corticosteroids
* No other malignant disease within the past 5 years except basalioma
* No functional iron deficiency (i.e., transferrin saturation < 20%) that cannot be treated with iron supplementation
* No other serious illness or medical condition

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 months since prior recombinant human epoetin alfa or any other erythropoiesis-stimulating drug

Chemotherapy

* At least 3 weeks since prior estramustine

Endocrine therapy

* See Disease Characteristics
* At least 3 weeks since prior antiandrogen treatment
* Concurrent chemical castration with LHRH allowed provided patient has begun treatment prior to study entry

  * No initiation of chemical castration therapy during study treatment

Radiotherapy

* No prior radiotherapy to > 25% of bone marrow
* No prior radioisotope therapy
* Concurrent local palliative radiotherapy for pain allowed

Surgery

* See Disease Characteristics
* At least 4 weeks since prior surgery

Other

* No other prior cytostatic treatment
* Concurrent bisphosphonates allowed provided patient has begun treatment prior to study entry

  * No initiation of bisphosphonates during study treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF)

SECONDARY OUTCOMES:
Quality of life every 6 weeks until TTF
Safety
Overall survival
Response rate
Use of epoetin beta

CONTACTS AND LOCATIONS:
Overall Officials: Pirkko Kellokumpu-Lehtinen, Principal Investigator — Tampere University Hospital
Locations (19):
- Finland (9):
  - Helsinki University Central Hospital, Helsinki
  - Kainuu Central Hospital, Kajaani
  - Keski-Pohjanmaa Central Hospital, Kokkola
  - Kymenlaakso Central Hospital, Kotka
  - Tampere University Hospital, Lahti
  - Oulu University Hospital, Oulu
  - Satakunta Central Hospital, Pori
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- Ireland (8):
  - Bons Secours Hospital, Cork
  - Mercy University Hospital, Cork
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Galway University Hospital, Galway
  - Mid-Western Cancer Centre at Mid-Western Regional Hospital, Limerick
- Sweden (2):
  - Karlstad Central Hospital, Karlstad
  - Karolinska University Hospital - Solna, Stockholm

REFERENCES:
- [Derived] Kellokumpu-Lehtinen PL, Harmenberg U, Joensuu T, McDermott R, Hervonen P, Ginman C, Luukkaa M, Nyandoto P, Hemminki A, Nilsson S, McCaffrey J, Asola R, Turpeenniemi-Hujanen T, Laestadius F, Tasmuth T, Sandberg K, Keane M, Lehtinen I, Luukkaala T, Joensuu H; PROSTY study group. 2-Weekly versus 3-weekly docetaxel to treat castration-resistant advanced prostate cancer: a randomised, phase 3 trial. Lancet Oncol. 2013 Feb;14(2):117-24. doi: 10.1016/S1470-2045(12)70537-5. Epub 2013 Jan 4. PMID 23294853
- [Derived] Hervonen P, Joensuu H, Joensuu T, Ginman C, McDermott R, Harmenberg U, Nyandoto P, Luukkaala T, Hemminki A, Zaitsev I, Heikkinen M, Nilsson S, Luukkaa M, Lehtinen I, Kellokumpu-Lehtinen PL. Biweekly docetaxel is better tolerated than conventional three-weekly dosing for advanced hormone-refractory prostate cancer. Anticancer Res. 2012 Mar;32(3):953-6. PMID 22399616